CLINICAL TRIAL: NCT00646542
Title: A Multi-center, Randomized, Double-blind Clinical Trial to Evaluate the Safety and Tolerability of 24 Weeks Treatment With (50 mg qd) Versus Placebo in Patients With Type 2 Diabetes and Moderate or Severe Renal Insufficiency
Brief Title: Safety and Tolerability of Vildagliptin Versus Placebo in Patients With Type 2 Diabetes and Moderate or Severe Renal Insufficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAF237A23137
Record Dates: First submitted 2008-03-24; First posted 2008-03-28 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes, vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Vildagliptin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin
  Other Names: Galvus
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This clinical trial is designed to provide additional information on the safety and tolerability of vildagliptin (50 mg once daily (qd)) when used in patients with type 2 diabetes mellitus (T2DM) and moderate or severe renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* History T2DM
* Moderate or Severe Renal Impairment

Exclusion Criteria:

* Glucose > 270 mg/dL (>15 mmol/L)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2005-03; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability in patients with T2DM and moderate or severe renal insufficiency over 24 weeks of treatment | 24 weeks

SECONDARY OUTCOMES:
To assess concentration levels of vildagliptin and its metabolites in patients with T2DM and moderate or severe renal insufficiency. | 24 weeks
To explore the efficacy of vildagliptin (50 mg qd) versus placebo in patients with T2DM and moderate or severe renal insufficiency. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (12):
- Buenos Aires, Argentina
- Heidelberg Heights, Australia
- Winnipeg, Canada
- Cartago, Costa Rica
- Tampere, Finland
- Angers, France
- Dormagen, Germany
- Chennai, India
- Oslo, Norway
- Saint Petersburg, Russia
- Alicante, Spain
- Lund, Sweden

REFERENCES:
- See also: Results for CLAF237A23137 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4598